CLINICAL TRIAL: NCT03634280
Title: Comparison of the Efficacy of Kinesio Taping and Splinting in Acute Treatment of Ankle Ligament Injuries
Brief Title: Efficacy of Kinesio Taping and Splinting in Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018.05.1.02.045
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Ankle Sprains
Keywords: Ankle Sprains; Kinesio Tape; Splint
MeSH Terms: conditions — Ankle Injuries | interventions — Splints

STUDY DESIGN:
Intervention Model Description: The patients were randomised using randomisation software and divided into two groups each comprising 120 patients. Tape and splint were kept on the patients for 5 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splinting (Placebo Comparator): Splinting was applied to the patients' ankle in the second group(n=120). Splint were kept on the patients for 5 days for 23 hours a day. In patients in the splint group, 16-18 layers of cotton gauze (15-cm cast gauze) were applied from the tip of the toes to the beginning of the fibula. Following the gauze application, short leg splint application was performed in a neutral ankle position.
  Interventions: Other: Kinesio taping
- Kinesio taping (Experimental): In this study, Kinesio Tape Tex Gold® kinesio tape over lateral ankle (5cm*5m) is used. 120 participants were taped for a lateral ankle sprain. 50-mm wide and 0.5-mm thick KT was applied to the tendinomuscular meridian around the ankle with three I-shaped tapes. Initially, one I-shaped tape was applied along the course of the tibialis anterior muscle, and another I-shaped tape was then applied to the peroneus longus and brevis muscles. The third I-shaped tape was applied from the abductor digiti minimi muscle and wrapped around the ankle in a figure-of-eight shape to the abductor hallucis muscle, surrounding the ankle over the medial and lateral malleoli. The tape was applied to the skin by applying zero tension, and skin problems were avoided.
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Other: Kinesio taping — In patients in the splint group, 16-18 layers of cotton gauze (15-cm cast gauze) were applied from the tip of the toes to the beginning of the fibula. Following the gauze application, short leg splint application was performed in a neutral ankle position.
  Other Names: Splinting

SUMMARY:
Question:Does kinesiotaping(KT) reduce oedema, pain, disability and increase range of joint motion on patients with acute ankle ligament injuries? Design:Two-group, randomised, controlled trial with blinded assessors. Participants:This study included 240 patients with acute ankle sprain.The patients were randomised using randomisation software and divided into two groups each comprising 120 patients.

Intervention:Tape and splint were kept on the patients for 5 days. Outcome measures:The following parameters were evaluated before and after treatment: circumference measurement for severity of oedema(metatarsophalangeal joint,ankle circumference,5cm above the ankle,10cm above the ankle),visual analog scale(VAS) pain score,range of motion(ROM) for the ankle with goniometer and disability level via the Foot Function Index (FFI).

DETAILED DESCRIPTION:
This study included 240 patients with acute ankle sprain admitted to the Emergency Department of Bağcılar Training and Research Hospital. Before initiating the study, approval of the Bağcılar Training and Research Hospital Clinical Investigations Ethics Committee was obtained with a decree number of 2018.05.1.02.045 dated 11/05/2018. The patients were randomised using randomisation software and divided into two groups each comprising 120 patients. Kinesio taping (KT) was applied to the patients in the first group, and splinting was applied to the patients in the second group. Tape and splint were kept on the patients for 5 days. Study inclusion criteria were age older than 18 years, presence of ankle sprain without osseous pathology and injury having occurred within the last 72 h. Exclusion criteria were the presence of fracture, open wound, motor or sensory deficits associated with injury, systemic oedema in the lower extremities related to the heart or kidney, venous diseases and past surgery.

The following parameters were evaluated before and after treatment: circumference measurement for severity of oedema (metatarsophalangeal joint, ankle circumference, 5 cm above the ankle, 10 cm above the ankle), VAS pain score, flexion, extension, inversion and eversion range of motion for the ankle with goniometer and disability level via the Foot Function Index (FFI).

The FFI is a widely used, self-administered instrument developed to measure the effects of foot pathologies on pain, disability and activity restriction. Turkish validity and reliability studies of FFI have been previously conducted. The FFI consists of 23 items assessed for three subscales: pain, disability and activity restriction. The pain subscale, which includes nine items, measures the level of foot pain in various situations, whereas the disability subscale, which includes nine items, identifies the degree of difficulty in performing various functional activities due to foot problems. The activity restriction subscale, which includes five items, is used to assess activity restriction due to foot problems. Patients score all items using a VAS, taking into account their foot condition 1 week earlier. To calculate subscale and total scale scores, the score of each item is summed, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability and activity restriction. If the patient is unable to perform activities, such as walking barefoot or using an orthosis, this item may be marked as not valid and removed from the total if possible.

Intervention KT application: 50-mm wide and 0.5-mm thick KT was applied to the tendinomuscular meridian around the ankle with three I-shaped tapes. Initially, one I-shaped tape was applied along the course of the tibialis anterior muscle, and another I-shaped tape was then applied to the peroneus longus and brevis muscles. The third I-shaped tape was applied from the abductor digiti minimi muscle and wrapped around the ankle in a figure-of-eight shape to the abductor hallucis muscle, surrounding the ankle over the medial and lateral malleoli. The tape was applied to the skin by applying zero tension, and skin problems were avoided.

In patients in the splint group, 16-18 layers of cotton gauze (15-cm cast gauze) were applied from the tip of the toes to the beginning of the fibula. Following the gauze application, short leg splint application was performed in a neutral ankle position.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Presence of ankle sprain without osseous pathology
* Injury having occurred within the last 72 h

Exclusion Criteria:

* Presence of fracture, open wound
* Motor or sensory deficits associated with injury
* Systemic oedema in the lower extremities related to the heart or kidney, venous diseases
* Past surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Disability | 5 minutes
  Foot Function Index: The FFI is designed to measure both current state, defined as the past week, and change in status. It consists of 23 items grouped into three sub-scales. Because the FFI was developed for use with a predominately elderly outpatient population, it was designed to be both short and simple. The number of items was minimized to reflect this consideration. The sub-scales were formed to provide information on three unique aspects of function-foot pain, disability and activity limitation-as they related to foot pathology. A score is derived for each item by dividing the attached horizontal line into 10 equal segments and assigning a number ranging from 0 to 9 to each segment. To obtain a sub-scale score, the item scores for a sub-scale are totaled and then divided by the maximum total possible for all of the sub-scale items which the patient indicated were applicable.

SECONDARY OUTCOMES:
Oedema | 3 minutes
  Circumference measurement for severity of oedema(metatarsophalangeal joint,ankle circumference,5cm above the ankle,10cm above the ankle)
Pain of ankle | 1 minute
  Visual analog scale
Range of motion | 3 minutes
  Range of motion for the ankle with goniometer

CONTACTS AND LOCATIONS:
Overall Officials: TOMRIS DUYMAZ, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided